CLINICAL TRIAL: NCT00323037
Title: A Multicenter,Randomized, Double Blind, Double Dummy, Parallel Group Study to Compare Effects of Coreg CR and Coreg IR on Left Ventricular End Systolic Volume Index in Subjects With Stable Chronic Heart Failure
Brief Title: A Study to Compare the Effects of Coreg CR and Coreg IR on Heart Function in Subjects With Stable Chronic Heart Failure
Acronym: COMPARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CTI-1, LLC (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104852
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Results first posted 2009-03-13 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Congestive Heart Failure
Keywords: heart failure
MeSH Terms: conditions — Heart Failure | interventions — Carvedilol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: carvedilol immediate release
- 2 (Active Comparator)
  Interventions: Drug: carvedilol controlled release

INTERVENTIONS:
Drug: carvedilol controlled release — Carvedilol controlled release (10, 20, 40 or 80 mg) and placebo taken in the morning. Two placebos taken in the evening. A total of 4 pills will be taken PO daily.
  Other Names: Coreg CR
  Arms: 2
Drug: carvedilol immediate release — Carvedilol immediate release (3.125, 6.25, 12.5 or 25 mg) and placebo, taken PO, twice-daily.
  Other Names: Coreg; Coreg IR
  Arms: 1

SUMMARY:
The purpose of this study is to determine if Coreg CR is as effective as Coreg IR in improving heart function in subjects with stable chronic heart failure.

DETAILED DESCRIPTION:
Results of clinical trials have shown beta-blockers improve symptoms and left ventricular function, reduce hospitalizations and death in heart failure, and prolong survival [MERIT-HF, CIBIS-II, Packer, 1996]. Clinical guidelines mandate use of beta-blockers in treatment of subjects with heart failure.

Carvedilol (Coreg IR) is a multiple action adrenergic receptor blocker with alpha 1, beta 1 and beta 2 receptor blockade properties. The beta-adrenergic properties are non-selective for beta 1 and beta 2 adrenergic receptors. Coreg IR, administered twice daily, is marketed in the United States for long term treatment of mild-moderate hypertension, mild to severe heart failure and subjects surviving an acute myocardial infarction with left ventricular dysfunction with or without symptomatic heart failure.

Coreg IR significantly reduces all cause mortality and the need for cardiovascular hospitalization [Packer, 1996a; Packer, 1996b; Colucci, 1996; Cohn, 1997; Olsen, 1995; Sharpe 1997]. The effect of Coreg is dose dependent [Bristow, 1996]. In subjects treated long term after an acute myocardial infarction (MI) complicated by left ventricular systolic dysfunction, Coreg IR reduced the frequency of all-cause and cardiovascular mortality, and recurrent non-fatal MIs. These beneficial effects are additional to those of evidence-based treatments for acute MI, including ACE inhibitors [Dargie, 2001].

Left Ventricular End Systolic Volume Index (LVESVI) is an important measure of ventricular function and remodeling in the evaluation of heart failure. In controlled clinical trials, Coreg IR, administered twice daily, has reduced LVESVI in subjects with ischemic heart failure. An echocardiography substudy of the Australia-New Zealand Trial [Doughty, 1997], evaluated left ventricular remodeling in 123 subjects with ischemic heart failure with an LVEF < 45 randomized to carvedilol or placebo. The LVESVI was reduced by 6.2 + 1.6 ml/m2 after 6 months and 8.7 + 2.6 ml/m2 after 12 months of carvedilol therapy compared to the placebo treated subjects. Metra et al [Metra, 2000] observed the favorable effects of carvedilol compared with metoprolol on LVEF, LV stroke volume, and pulmonary artery pressure despite similar effects on cardiovascular outcome. Both groups also showed significant decreases in LV systolic volume. Doughty et al [Doughty, 2004] observed the favorable effects of carvedilol on LV remodeling, with improved LV end-systolic volume and ejection fraction, after 6 months of treatment.

Carvedilol phosphate CR (Coreg CR) is an approved, modified release, once-daily formulation of carvedilol that is hoped to provide an advance in patient care through improved compliance with prescribed dose.

The clinical experience with various formulations of Coreg CR is limited to eight single dose studies in healthy subjects and one repeated dose study in subjects with hypertension. In total 230, adult subjects have received at least one dose of Coreg IR or one of several CR formulations across nine studies. The subjects ranged in age from 18 to 63 years; 62% were male and 69% were white. The various formulations of Coreg CR capsules were safe and well tolerated in single dose pharmacokinetic studies in doses ranging from 6.25 to 60 mg in healthy subjects. The most common adverse events were headache, dizziness and orthostatic hypotension and are all known adverse events following administration of Coreg IR [GSK Study 386, 388, 399, 400, 402, 907].

This study will be the first controlled clinical study investigating the efficacy of treatment with Coreg CR formulation [Coreg CR filled with 7.5 mg of carvedilol phosphate immediate release (IRp) microparticles, 22.5 mg of carvedilol phosphate Micropump IIa MR microparticles, and 30 mg of carvedilol phosphate Micropump IIc MR microparticles] compared to Coreg IR evaluating LVESVI in subjects with stable chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female
* At least 18 years of age at the time informed consent is signed
* Stable, chronic, mild to severe heart failure as defined as subjects with symptoms of heart failure who do not require IV diuretics, inotropes, or vasodilators or those that require support with a left ventricular assist device
* Angiotensin converting enzyme inhibitors or angiotensin receptor blockers should be prescribed to all patients with HF due to LV systolic dysfunction with reduced LVEF unless contraindicated or intolerant to use
* At screening, subject has an LVEF < 40 as measured by 2-D echocardiography
* Willing to provide written informed consent

Exclusion Criteria:

* On beta-blocker therapy for greater than 42 days prior to consent
* Acute ischemic coronary event or coronary revascularization (PTCA, CABG, thrombolysis) within 1 week of screening echocardiography
* Scheduled or expected to be scheduled coronary revascularization within 4 weeks
* Unstable angina (angina characterized by sudden changes in the severity or length of angina attacks or a decrease in level of exertion that precipitates an episode
* Uncorrected primary obstructive or severe regurgitant valvular disease, nondilated (restrictive) or hypertrophic cardiomyopathies
* Uncontrolled ventricular arrhythmias (symptomatic or sustained ventricular arrhythmias not controlled with antiarrhythmic therapy or an implantable defibrillator)
* Current treatment of calcium channel blockers except for long acting dihydropyridines
* Current treatment on any Class I or III antiarrhythmic, except amiodarone
* History of sick sinus syndrome unless a pacemaker is in place
* Second or third degree heart block unless a pacemaker is in place
* Current clinical evidence of obstructive pulmonary disease (e.g., asthma or bronchitis) requiring inhaled or oral bronchodilator or steroid therapy; or having a history of bronchospastic disease not undergoing active therapy in whom, in the investigator's opinion, treatment with study medication could provoke bronchospasm
* Expected biventricular pacemaker placement within 8 months of enrollment
* Resting systolic blood pressure <90 mmHg (based on the average of 3 readings
* Resting heart rate <50 beats per minute (bpm) (based on the average of 3 readings)
* Current decompensated heart failure
* Elevated liver enzymes (i.e., ALT or AST levels greater than 3 times upper limit of normal)
* History of drug sensitivity or allergic reaction to alpha or beta-blockers
* Contraindication or intolerance to beta-blockers
* Pregnant or lactating women and women planning to become pregnant. NOTE: Female subjects must be post-menopausal (i.e., no menstrual period for a minimum of 6 months prior to screening), surgically sterilized, using a double barrier method contraceptive, or using Depo-Provera or implanted contraceptives for at least one month prior to screening and agree to continue to use the same contraceptive method throughout the study.
* Use of an investigational drug within 30 days of enrollment
* Participation in an investigational device trial within 30 days of enrollment
* Known drug or alcohol abuse 1 year prior to enrollment
* In the opinion of the investigator the subject is known to be noncompliant with prescribed medication regimen
* Has any systemic disease, including cancer, with reduced life expectancy (<12 months)
* Has a history of psychological illness/condition that interferes with ability to understand or complete requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Greenberg, MD, Study Chair
Locations (75):
- United States (75):
  - Cardiology Associates, Mobile, Alabama
  - Mobile Heart Specialists, Mobile, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Scottsdale Cardiovascular Research Institute, Scottsdale, Arizona
  - South West Heart, Tucson, Arizona
  - Inland Heart Doctors Medical Group, Corona, California
  - Rancho Los Amigos USC, Downey, California
  - William Bowden, DO Private Practice, Healdsburg, California
  - Merced Heart Associates, Merced, California
  - Sutter Memorial Hospital, Sacramento, California
  - Southern California Cardiology Medical Group, Inc., San Diego, California
  - Medvin Clinical Research, Van Nuys, California
  - Aurora Denver Cardiology Associates, Denver, Colorado
  - Medical Center of the Rockies Foundation, Loveland, Colorado
  - Bay Area Cardiology, Brandon, Florida
  - Clearwater Cardiovascular and Interventional Consultants, Clearwater, Florida
  - White-Wilson Medical Center, PA, Fort Walton Beach, Florida
  - South Florida International Cardiology Consultants, Inc., Miami, Florida
  - Palm Beach Cardiology, Palm Beach Gardens, Florida
  - Cardiac Disease Specialists, PC, Atlanta, Georgia
  - Harbin Clinic, Rome, Georgia
  - North Shore Cardiovascular Research Consortium, Bannockburn, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Illinois Heart and Vascular, Hinsdale, Illinois
  - HeartCare Midwest, Peoria, Illinois
  - Rockford Cardiology Research Foundation, Rockford, Illinois
  - Prairie Cardiovascular Consultants, Springfield, Illinois
  - The Care Group LLC, Indianapolis, Indiana
  - River Cities Cardiology, Jeffersonville, Indiana
  - Iowa Heart Center, West Des Moines, Iowa
  - Mid-America Cardiology, Kansas City, Kansas
  - Via Christi Research, Inc., Wichita, Kansas
  - Comprehensive Cardiology Associates, Florence, Kentucky
  - Cardiovascular Associates, Louisville, Kentucky
  - Louisville Cardiology Medical Group, Louisville, Kentucky
  - One Heart, LLC, Baltimore, Maryland
  - Minnesota Heart Clinic, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Regions Hospital Cardiology Research, Saint Paul, Minnesota
  - St. Paul Cardiology, Saint Paul, Minnesota
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Rocky Mountain Heart & Lung, Kalispell, Montana
  - Diagnostic and Clinical Cardiology, West Orange, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Albany Associates in Cardiology, Albany, New York
  - Buffalo Heart Group, LLP, Buffalo, New York
  - Long Island Heart Associates, Mineola, New York
  - New York Cardiovascular Associates, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - South Bay Cardiovascular Associates, West Islip, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Sterling Research Group Ltd., Cincinnati, Ohio
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - University Hospital, Cincinnati, Ohio
  - Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Samaritan Cardiology, Corvallis, Oregon
  - Blair Medical Associates, Altoona, Pennsylvania
  - Tri-State Medical Group, Beaver, Pennsylvania
  - Central Bucks Specialists, Doylestown, Pennsylvania
  - Cardiology Consultants of Philadelphia, Philadelphia, Pennsylvania
  - Mid State Medical Service, Philipsburg, Pennsylvania
  - Buxmont Cardiology Associates, PC, Sellersville, Pennsylvania
  - Rhode Island Heart Failure Center, Providence, Rhode Island
  - Charleston Cardiology, Charleston, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - Heart Specialists, Friendswood, Texas
  - Texas Cardiac Center, Lubbock, Texas
  - Intermountain Medical Center, Murray, Utah
  - Heart Center, Salt Lake City, Utah
  - Winchester Medical Center, Winchester, Virginia
  - Luther Midelfort Mayo Health Systems, Eau Claire, Wisconsin
  - Green Bay HeartCare, Green Bay, Wisconsin

REFERENCES:
- [Background] Effect of metoprolol CR/XL in chronic heart failure: Metoprolol CR/XL Randomised Intervention Trial in Congestive Heart Failure (MERIT-HF). Lancet. 1999 Jun 12;353(9169):2001-7. PMID 10376614
- [Background] The Cardiac Insufficiency Bisoprolol Study II (CIBIS-II): a randomised trial. Lancet. 1999 Jan 2;353(9146):9-13. PMID 10023943
- [Background] Packer M, Colucci WS, Sackner-Bernstein JD, Liang CS, Goldscher DA, Freeman I, Kukin ML, Kinhal V, Udelson JE, Klapholz M, Gottlieb SS, Pearle D, Cody RJ, Gregory JJ, Kantrowitz NE, LeJemtel TH, Young ST, Lukas MA, Shusterman NH. Double-blind, placebo-controlled study of the effects of carvedilol in patients with moderate to severe heart failure. The PRECISE Trial. Prospective Randomized Evaluation of Carvedilol on Symptoms and Exercise. Circulation. 1996 Dec 1;94(11):2793-9. doi: 10.1161/01.cir.94.11.2793. PMID 8941104
- [Background] Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, Shusterman NH. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996 May 23;334(21):1349-55. doi: 10.1056/NEJM199605233342101. PMID 8614419
- [Background] Colucci WS, Packer M, Bristow MR, Gilbert EM, Cohn JN, Fowler MB, Krueger SK, Hershberger R, Uretsky BF, Bowers JA, Sackner-Bernstein JD, Young ST, Holcslaw TL, Lukas MA. Carvedilol inhibits clinical progression in patients with mild symptoms of heart failure. US Carvedilol Heart Failure Study Group. Circulation. 1996 Dec 1;94(11):2800-6. doi: 10.1161/01.cir.94.11.2800. PMID 8941105
- [Background] Cohn JN, Fowler MB, Bristow MR, Colucci WS, Gilbert EM, Kinhal V, Krueger SK, Lejemtel T, Narahara KA, Packer M, Young ST, Holcslaw TL, Lukas MA. Safety and efficacy of carvedilol in severe heart failure. The U.S. Carvedilol Heart Failure Study Group. J Card Fail. 1997 Sep;3(3):173-9. doi: 10.1016/s1071-9164(97)90013-0. PMID 9330125
- [Background] Olsen SL, Gilbert EM, Renlund DG, Taylor DO, Yanowitz FD, Bristow MR. Carvedilol improves left ventricular function and symptoms in chronic heart failure: a double-blind randomized study. J Am Coll Cardiol. 1995 May;25(6):1225-31. doi: 10.1016/0735-1097(95)00012-S. PMID 7722114
- [Background] Randomised, placebo-controlled trial of carvedilol in patients with congestive heart failure due to ischaemic heart disease. Australia/New Zealand Heart Failure Research Collaborative Group. Lancet. 1997 Feb 8;349(9049):375-80. PMID 9033462
- [Background] Bristow MR, Gilbert EM, Abraham WT, Adams KF, Fowler MB, Hershberger RE, Kubo SH, Narahara KA, Ingersoll H, Krueger S, Young S, Shusterman N. Carvedilol produces dose-related improvements in left ventricular function and survival in subjects with chronic heart failure. MOCHA Investigators. Circulation. 1996 Dec 1;94(11):2807-16. doi: 10.1161/01.cir.94.11.2807. PMID 8941106
- [Background] Dargie HJ. Effect of carvedilol on outcome after myocardial infarction in patients with left-ventricular dysfunction: the CAPRICORN randomised trial. Lancet. 2001 May 5;357(9266):1385-90. doi: 10.1016/s0140-6736(00)04560-8. PMID 11356434
- [Background] Doughty RN, Whalley GA, Walsh HA, Gamble GD, Lopez-Sendon J, Sharpe N; CAPRICORN Echo Substudy Investigators. Effects of carvedilol on left ventricular remodeling after acute myocardial infarction: the CAPRICORN Echo Substudy. Circulation. 2004 Jan 20;109(2):201-6. doi: 10.1161/01.CIR.0000108928.25690.94. Epub 2004 Jan 5. PMID 14707020
- [Background] Doughty RN, Whalley GA, Gamble G, MacMahon S, Sharpe N. Left ventricular remodeling with carvedilol in patients with congestive heart failure due to ischemic heart disease. Australia-New Zealand Heart Failure Research Collaborative Group. J Am Coll Cardiol. 1997 Apr;29(5):1060-6. doi: 10.1016/s0735-1097(97)00012-0. PMID 9120160
- [Background] Greenberg BH, Mehra M, Teerlink JR, Ordronneau P, McCollum D, Gilbert EM. COMPARE: comparison of the effects of carvedilol CR and carvedilol IR on left ventricular ejection fraction in patients with heart failure. Am J Cardiol. 2006 Oct 2;98(7A):53L-59L. doi: 10.1016/j.amjcard.2006.08.003. Epub 2006 Aug 28. PMID 17023233

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from April 2006 until August 2007.
Period: Overall Study
Arm/Group | Coreg Immediate Release | Coreg Controlled Release
Started | 165 (Number randomized) | 153 (Number randomized)
Completed | 132 | 126
Not Completed | 33 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coreg Immediate Release | Coreg Controlled Release | Total
Number analyzed (Participants) | 165 | 153 | 318
Age, Customized [Number; unit: participants]
  < 65 years | 117 | 110 | 227
  65<=Age<75 | 27 | 21 | 48
  Age>=75 years | 21 | 22 | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 45 | 97
  Male | 113 | 108 | 221

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Left Ventricular End Systolic Volume Index (LVESVI) Characterized by 2-D Echocardiography
Description: Maintenance Visit 3 minus Baseline. Maintenance Visit 3 occurred 24 weeks after entry into the maintenance period. The maintenance period started after completion of a titration period of variable duration.
Time Frame: 24 weeks after entry into the maintenance period
Population: Analysis was performed on the modified intent to treat population (mITT), which were those subjects with both a Baseline and an evaluable End of Study echocardiogram.
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Coreg Immediate Release | Coreg Controlled Release
Number analyzed (Participants) | 128 | 125
mL/m^2 | -18.36 (18.84) | -20.81 (25.43)

2. Secondary Outcome: Change From Baseline in Left Ventricular Ejection Fraction (LVEF)
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 128 | 125
percentage of change | .08 (.10) | .08 (.10)

3. Secondary Outcome: Change From Baseline in Left Ventricular End Diastolic Volume (LVEDV)
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 128 | 125
percentage of change | -36.61 (46.27) | -42.22 (64.89)

4. Secondary Outcome: Change From Baseline in Left Ventricular End Systolic Volume (LVESV)
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 128 | 125
percentage of change | -36.61 (46.27) | -43.00 (53.49)

5. Secondary Outcome: Change From Baseline in Left Ventricular End Diastolic Volume Index (LVEDVI)
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 128 | 125
percentage of change | -18.29 (22.61) | -20.57 (31.28)

6. Secondary Outcome: Change From Baseline in Intraventricular Septal Thickness (IVST)
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 75 | 79
percentage of change | .08 (.26) | .05 (.26)

7. Secondary Outcome: Change From Baseline in Posterior Wall Thickness (PWT)
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 67 | 69
percentage of change | .07 (.23) | .05 (.23)

8. Secondary Outcome: Change From Baseline in Left Ventricular Mass (LVM)
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 59 | 55
percentage of change | 9.5 (113.43) | -9.29 (105.06)

9. Secondary Outcome: Change From Baseline in End Diastolic Dimension (EDD)
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 64 | 57
percentage of change | -0.33 (.97) | -0.36 (.95)

10. Secondary Outcome: Change From Baseline in End Systolic Dimension (ESD)
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 61 | 55
percentage of change | -0.76 (1.08) | -0.83 (1.14)

11. Secondary Outcome: Change From Baseline in Deceleration Time
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 92 | 95
percentage of change | 24.00 (91.71) | 53.37 (83.74)

12. Secondary Outcome: Change From Baseline in Early to Late Atrial Ratio (E:A Ratio)
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 84 | 86
percentage of change | -0.20 (0.70) | -0.45 (0.75)

13. Secondary Outcome: Change From Baseline in BNP Levels
Time Frame: 24 weeks after entry into the maintenance period
Population: modified intent to treat subjects
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 121 | 116
percentage of change | -0.88 (1.25) | -0.86 (1.16)

14. Secondary Outcome: Incidence of Hospitalizations
Time Frame: Up to 32 weeks (titration and maintenance phases)
Population: intent to treat subjects
Measure: Number; unit: participants in each treatment group
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 165 | 153
participants in each treatment group
  Hospitalization for Heart Failure | 6 | 6
  Hospitalization Due to Any Cause | 31 | 29
  Hospitalization or Death | 32 | 29

15. Secondary Outcome: Drug Dose Tolerability
Time Frame: Up to 32 weeks (titration and maintenance phases)
Population: intent to treat subjects
Measure: Number; unit: subjects in each treatment group
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 165 | 153
subjects in each treatment group
  Study Entry (10mg Coreg CR, 3.125mg Coreg IR) | 79 | 83
  Maintenance Entry (10mg Coreg CR, 3.125mg Coreg IR) | 0 | 0
  End of Study (10mg Coreg CR, 3.125mg Coreg IR) | 7 | 4
  Study Entry (20mg Coreg CR, 6.25mg Coreg IR) | 61 | 39
  Maintenance Entry (20mg Coreg CR, 6.25mg Coreg IR) | 13 | 9
  End of Study (20mg Coreg CR, 6.25mg Coreg IR) | 16 | 16
  Study Entry (40mg Coreg CR, 12.5mg Coreg IR) | 21 | 27
  Maintenance Entry (40mg Coreg CR, 12.5mg Coreg IR) | 12 | 16
  End of Study (40mg Coreg CR, 12.5mg Coreg IR) | 21 | 22
  Study Entry (80mg Coreg CR, 25mg Coreg IR) | 4 | 4
  Maintenance Entry (80mg Coreg CR, 25mg Coreg IR) | 116 | 114
  End of Study (80mg Coreg CR, 25mg Coreg IR) | 121 | 111

16. Secondary Outcome: Treatment Compliance
Time Frame: Up to 32 weeks (titration and maintenance phases)
Population: intent to treat subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 142 | 132
Participants
  <80% compliance | 4 | 6
  80%-120% | 138 | 126

17. Secondary Outcome: Safety and Tolerability of Coreg CR
Description: SAEs experienced
Time Frame: 24 weeks after entry into the maintenance phase (after unblinding)
Population: intent to treat
Measure: Number; unit: number of SAEs
Arm/Group | Carvedilol Immediate Release | Carvedilol Controlled Release
Number analyzed (Participants) | 27 | 27
number of SAEs | 40 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The publishing party will submit any proposed manuscript or publication to the sponsor for comment at least 60 days prior to its release. The publishing party will make every reasonable attempt to incorporate comments received from the sponsor, and will upon request remove any previously undisclosed confidential information, prior to publication or disclosure. There will be no publication or publicizing of individual site data or results prior to the multicenter publication.